CLINICAL TRIAL: NCT06827054
Title: Low-Dose Psilocybin Therapy for Palliative Care Patients With Chronic Cancer Pain Requiring Opioids
Brief Title: Psilocybin With Psychotherapy for Improving Chronic Pain in Cancer Patients Requiring Opioids
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I-3914823; NCI-2024-10761 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3914823 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-01-22; First posted 2025-02-14 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Specimen Handling; Interviews as Topic; Psilocybin; Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Supportive care (psychotherapy, psilocybin) (Experimental): Patients attend two preparatory psychotherapy sessions. Patients then receive psilocybin PO BIW for 4 weeks (8 doses total) in the absence of unacceptable toxicity and attend three integration psychotherapy sessions over 1.5 hours each during psilocybin dosing sessions 2, 4, and 6. Patients may optionally attend additional psychotherapy sessions as needed during follow-up. Additionally, patients undergo fMRI and collection of blood and urine samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Functional Magnetic Resonance Imaging; Other: Interview; Drug: Psilocybine; Behavioral: Psychotherapy; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and urine samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Functional Magnetic Resonance Imaging — Undergo fMRI
  Other Names: fMRI; Functional MRI
Other: Interview — Ancillary studies
Drug: Psilocybine — Given PO
  Other Names: CY-39; Indocybin; Psilocybin
Behavioral: Psychotherapy — Attend psychotherapy sessions
  Other Names: talk therapy
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies whether psilocybin with psychotherapy is safe and if it works for improving chronic pain in cancer patients who require opioids to manage their pain. Psilocybin is taken from the mushroom Psilocybe mexicana. Psilocybin acts on the brain to cause hallucinations (sights, sounds, smells, tastes, or touches that a person believes to be real but are not real). This may impact a patient's "total pain", a view that accounts for the psychological, spiritual, and social factors that contribute to their experience of pain. Psychotherapy uses methods such as discussion, listening, and counseling to help patients change the way they react to environmental triggers that may cause a negative reaction. Giving psilocybin with psychotherapy may be safe and helpful for improving chronic pain in cancer patients who require opioids to manage their pain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety, tolerability, and feasibility of low dose psilocybin therapy in patients with chronic cancer pain who require opioids.

SECONDARY OBJECTIVE:

I. To obtain preliminary evidence for efficacy of low dose psilocybin therapy in reducing pain and opioid requirement in participants with chronic cancer pain.

EXPLORATORY OBJECTIVES:

I. To evaluate potential mechanisms of action for psilocybin in pain control, including its effects on resting brain network activity, inflammation, and psychological changes processes.

II. To obtain preliminary evidence for efficacy of psilocybin therapy on additional outcomes related to pain control, physical function, and opioid requirement in participants with chronic cancer pain.

III. To obtain preliminary evidence for efficacy of low dose psilocybin therapy in alleviating psychological symptoms associated with chronic cancer pain.

IV. To evaluate potential mechanisms of action for low dose psilocybin therapy in pain control, including its effects on the following: resting brain network activity, inflammation, psychological processes and psychedelic effects.

OUTLINE:

Patients attend two preparatory psychotherapy sessions. Patients then receive psilocybin orally (PO) twice a week (BIW) for 4 weeks (8 doses total) in the absence of unacceptable toxicity and attend three integration psychotherapy sessions over 1.5 hours each during psilocybin dosing sessions 2, 4, and 6. Patients may optionally attend additional psychotherapy sessions as needed during follow-up. Additionally, patients undergo functional magnetic resonance imaging (fMRI) and collection of blood and urine samples throughout the study.

After completion of study intervention, patients are followed up at days 28-34, 56, and 84.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years old
* Diagnosis of active cancer, any stage
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Estimated prognosis of ≥ 3 months at the time of enrollment, determined by participant's primary oncologist or palliative physician
* Diagnosis of moderate to severe pain (reported average pain score ≥ 4 on the 11-point Numerical Rating Scale) that is chronic (≥ 3 months) and secondary to cancer or cancer treatment
* Pain regimen has been escalated to opioid therapy

  * Participants must be on stable pain regimen for at least one month prior, with no intention to adjust pain regimen during the study period
* Participants must be ≥ 4 weeks beyond treatments/procedures that, in the opinion of the study physician, would significantly affect outcomes related to pain and physical function (e.g., surgery or radiation). Participants may otherwise receive cancer-directed treatment throughout the study period
* Have no known procedures/treatments scheduled in advance that would prohibit patient from completing or significantly delaying completion of the study

  * The participant has no vacations or plans to be out of town during their study enrollment
* Participants must not plan for additional treatments/procedures that, in the opinion of the study physician, would significantly affect outcomes related to pain and physical function (e.g., surgery or radiation) for ≥ 4 weeks following psilocybin treatment initiation. Participants may otherwise receive cancer-directed treatment throughout the study period
* No use of other illicit substances (excluding cannabis) within the past year based on self-report at screening and routine urine toxicology screen
* Participants must be able to read, write, and speak English
* Participants must be able to swallow pills
* Agree to refrain from using any unprescribed psychoactive drugs, including alcoholic beverages, ≤ 24 hours of before each psilocybin administration. Exceptions include:

  * Daily use of caffeine or nicotine
  * Prescribed benzodiazepine medications and non-benzodiazepine sleeping medications will be allowed to continue through the study period for participants who have been on a stable dose of such a medicine for ≥ 6 weeks prior to screening
* Participants using cannabis, including legal cannabis, for any purpose must agree to refrain from use beginning at two weeks before dosing and one week following completion of dosing (7-8 weeks total, dependent on frequency of prior use)

  * Participants will not be withdrawn from the trial for a positive cannabis result during the initial screening drug test. However, participants who test positive for cannabis at the second drug test on visit 10 will be withdrawn from the trial
* Participants must agree to be driven home after each experimental session and not drive or operate heavy machinery ≤ 16 hours of ingesting psilocybin
* Participants must provide an emergency contact (relative, spouse, close friend, or other support person) willing and able to be reached by the investigators if the participant is unreachable by study staff or in an emergency
* The participant agrees to take part in all study procedures, including the assessments, psychological evaluations, and dosing day requirements
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Participants who are pregnant or breast-feeding
* Participants of childbearing potential who decline to use a highly effective dual contraceptive method for the duration of the study
* Participants with a condition impairing oral intake or digestive absorption
* Cognitive impairment as defined by Montreal Cognitive Assessment (MOCA) score < 23
* Medical conditions or serious abnormalities of complete blood count, chemistries, or electrocardiography (ECG) that in the opinion of the study physician would preclude safe participation in the trial. Some examples include: congestive heart failure, valvular heart disease, recent acute myocardial infarction or evidence of ischemia, clinically significant arrhythmias (e.g., ventricular fibrillation, torsades) or clinically significant ECG abnormality (e.g. corrected QT interval using Fridericia's Correction Formula [QTcF] interval > 450 in males and > 470 in females), uncontrolled hypertension (systolic blood pressure [BP] ≥ 140 or diastolic BP ≥ 90 on three separate occasions), congenital long QT syndrome, renal dysfunction (i.e. creatinine clearance [CrCl] < 40 mL/min), liver cirrhosis or hepatic dysfunction (indicated by gamma-glutamyltransferase [GGT], aspartate aminotransferase [AST], or alanine aminotransferase [ALT] > 3 x ULN [upper limit of norm] or total bilirubin [bili] > 3.0 mg/dl, or Child Pugh over class C), paraneoplastic syndrome, respiratory failure, dementia, delirium, known cerebral aneurysm, seizure disorder, stroke/transient ischemic attack (TIA) in past year, cancer with known central nervous system (CNS) involvement, previously treated brain metastasis, or other major CNS disease
* Participants who have a personal history of, or a current diagnosis of the following: primary psychotic disorder, major depressive disorder with psychotic features, bipolar affective disorder type 1 or history of or current dissociative identity disorder
* Participants who have an ongoing substance use disorder (defined as active in the past year)
* Participants with first-degree relatives with schizophrenia or bipolar disorder may be eligible depending on their age and personal and family psychiatric history. The decision will be made by the principal investigator and study psychiatrist or on-call psychiatric provider based on risk assessment
* Active suicidal behavior (interrupted or aborted attempt; preparatory acts) as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) connotating either passive or active suicidal intent; OR one of the following:

  * History of suicide attempt(s) within the past year (≤ 365 days)
  * Have any suicidal ideation or thoughts, in the opinion of the study physician or principal investigator (PI), that presents a serious risk of suicidal or self-injurious behavior
* Any contraindications to undergoing an fMRI scan, including having metal implants or metal fragments in the body
* Participants who have hypersensitivity to the ingredients of the IMP (Investigational Medicinal Product) listed below:

  * Indol alkaloids including psilocybin and psilocin
  * Constituents of Psilocybe cubensis including protein, fats, carbohydrates, ergosterols, beta-glucan, and polyphenols
  * Hydroxypropyl methylcellulose (HPMC) capsules
* Participants who are taking medications with significant potential to interact with study medications will be exclusionary if they cannot be tapered. The taper interval will be at least five times the half-life. These medications include the following:

  * Selective serotonin reuptake inhibitors (SSRIs)
  * Serotonin and norepinephrine reuptake inhibitors (SNRIs)
  * Tricyclic antidepressants (TCAs)
  * Efavirenz
  * Serotonin-acting dietary supplements (i.e., 5-hydroxy-tryptophan or St. John's wort)
  * Centrally acting serotonergic agents (e.g., monoamine oxidase [MAO] inhibitors)
  * Antipsychotics for a psychiatric disorder (e.g., first and second generation)

    * Antipsychotics that are utilized for nausea, insomnia, or other non-psychiatric condition will be permitted, but patients will be asked to refrain from use 8 hours prior to dosing sessions
  * Mood stabilizers (e.g., lithium, valproic acid)
  * Aldehyde dehydrogenase inhibitors (e.g., disulfiram)
  * Significant inhibitors of UGT 1A9 or UGT 1A10
* Use of serotonergic hallucinogens (e.g., psilocybin, lysergic acid diethylamine [LSD]) within the past 12 months or significant lifetime use (> 25 uses)
* Those with a history of prior violent and/or drug-related felonies
* Those currently incarcerated will be excluded
* Unwilling or unable to follow protocol requirements
* Any social circumstance which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-05-05 (Estimated); Study Completion 2027-05-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From start date of intervention to 30 days after the last intervention
  AE assessments will be performed at each treatment session and all subsequent in-person and virtual visits. This will be clinician-observed events. These evaluations will utilize the established Common Terminology Criteria for Adverse Events version 5.0. AEs will be summarized by attribution and grade using frequencies and relative frequencies, where the grade 3+ AE rate will be estimated with 90% credible regions obtained by Jeffrey's prior method. Additionally, a continual safety monitoring plan will be utilized to ensure study suspension should the AE rates exceed pre-defined thresholds.
Change in Vital signs | Up to baseline, dosing sessions 1 and 2 up to day 84
  Continuous Vital signs will be assessed and summarized by timepoint using the appropriate descriptive statistics. The change in these measures will be modeled as a function of time and a random subject effect using linear mixed models, where tests about the appropriate contrasts of model estimates will be used to identify significant changes relative to pre-treatment levels. All model assumptions will be verified graphically.
Incidence of clinically important changes in ICG parameters | At baseline and day 28
  To assess any changes in EKG records from baseline EKG to day 28 EKG
Change in risk for suicide | At baseline, dosing sessions 1, 2, 3, 5, and 7, and days 28, 56, and 84
  Will be assessed using the Columbia-Suicide Severity Rating Scale. Will be summarized by timepoint using the appropriate descriptive statistics. The change will be modeled as a function of time and a random subject effect using linear mixed models, where tests about the appropriate contrasts of model estimates will be used to identify significant changes relative to pre-treatment levels. All model assumptions will be verified graphically.
Change in cognitive function | At dosing sessions 1-3 and days 28, 56, and 84
  A Montreal Cognitive Assessment will be provided prior to the first dosing session, at two-hour intervals during the first two dosing sessions and subsequent dosing sessions if a dose reduction occurred, and once during subsequent visits.
Recruitment rate | Up to day 84
  Recruitment will be measured as a percentage of participants who were contacted for prescreening that were enrolled. Will be estimated with 90% credible regions obtained by Jeffrey's prior method.
Retention rate | Up to day 84
  Retention rate will be measured as a percentage of participants who enrolled that completed the trial, determined by completion of visit 19. Will be estimated with 90% credible regions obtained by Jeffrey's prior method.

SECONDARY OUTCOMES:
Change in average pain intensity | At baseline and days 3, 7, 28, 56, and 84
  The reported average pain will be assessed via the Brief Pain Inventory-Short Form, which includes multiple pain-related questions using an 11-point Numerical Rating Scale. A decrease by 30% or 2 points is regarded as clinically meaningful. Will be summarized by timepoint (baseline and by micro-dose session) using the appropriate descriptive statistics and graphical summaries. The log of each outcome will be modeled as a function of timepoint and a random subject effect using a linear mixed model. Tests about the appropriate contrasts of model estimates will be used to evaluate changes of interest. All model assumptions will be verified graphically.
Change in rescue opioid requirement | At baseline and days 3, 7, 28, 56, and 84
  Will be measured in Oral Morphine Equivalents. Will be assessed via participant self-report with medication log and further verified with pill count. Will be summarized by timepoint (baseline and by micro-dose session) using the appropriate descriptive statistics and graphical summaries. The log of each outcome will be modeled as a function of timepoint and a random subject effect using a linear mixed model. Tests about the appropriate contrasts of model estimates will be used to evaluate changes of interest. All model assumptions will be verified graphically.

CONTACTS AND LOCATIONS:
Overall Officials: William Alexander, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States